CLINICAL TRIAL: NCT03991923
Title: Non-ischemic Preservation of the Donor Heart in Heart Transplantation - a Randomized, Controlled, Multicenter Trial
Brief Title: Non-ischemic Preservation of the Donor Heart in Heart Transplantation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: XVIVO Perfusion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NIHP2019
Record Dates: First submitted 2019-06-04; First posted 2019-06-19 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Heart Transplantation
Keywords: Non Ischemic Heart Preservation (NIHP); Ischemic cold static storage of donor hearts (ICSS)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Non-ischemic heart preservation (NIHP) (Experimental): Continous cold cardioplegic perfusion of hearts
  Interventions: Device: XVIVO heart preservation devices
- Ischemic cold static storage (ICSS) (Active Comparator): Standard preservation technique
  Interventions: Device: Standard ICSS

INTERVENTIONS:
Device: XVIVO heart preservation devices — The intervention is to preserve hearts during transportation cold, cardioplegic and non-ischemic, with a high oncotic and hormone supplemented perfusate.
  Arms: Non-ischemic heart preservation (NIHP)
Device: Standard ICSS — Cold static preservation using standard preservation solution
  Arms: Ischemic cold static storage (ICSS)

SUMMARY:
The study intends to compare standard ischemic cold static storage (ICSS) of retrieved hearts intended to be transplanted, to non-ischemic heart preservation (NIHP) in a randomized clinical multicentre trial. The primary hypothesis is that the non-ischemic hypothermic cardioplegic preservation (NIHP) is safe and superior to ischemic cold static storage (ICSS) of donor hearts. The study will investigate the safety and superiority of the new methodology in terms of improved immediate and prolonged organ function in adult heart transplanted patients.

DETAILED DESCRIPTION:
This study will investigate if non-ischemic heart preservation (NIHP) with the XVIVO heart preservation devices could improve clinical outcome of patients receiving hearts after use of the technology compared to after use of standard cold ischemic preservation. This will be investigated in a European multicentre randomized controlled clinical trial. For technical reasons, blinding to the involved clinical personnel is not possible, however, biopsies will be blinded to study pathologists. The trial will include 202 recipients that have been randomized through their heart donor. The primary outcome of the study is a clinically relevant composite including graft survival, primary graft dysfunction, rejection and use of circulatory mechanical support, within 30 days and also including Cardiac Allograft Vasculopathy within 12 months. As secondary outcomes, molecular markers related to cardiac injury CKMB, ProBNP and TNI will be investigated as well as markers of the inflammatory response. Safety aspects such as effect on other organs and machine defects will also be monitored. The study population is adults, listed for heart transplantation and donors accepted as heart donors according to standard hospital procedures. Specific recipient exclusion criteria related to pre-transplant ECMO support, patients undergoing pre-transplant desensitization protocol, patients with Grown-Up Congenital Heart Disease, patients with severe kidney or liver dysfunction, patients with septicaemia, and patients diagnosed with Systemic Lupus Erythematous, sarcoidosis or amyloidosis are excluded. Cardiac death donors and donors with previous sternotomy are excluded. The study hypothesis is that NIHP better preserves the endothelium and myocyte function of the heart resulting in improved short- and medium-term recipient outcome, without inducing any new significant risks to the retrieved heart or the recipient. This is believed to be accomplished through continuous oxygenation of the heart via perfusion of the coronary arteries using an optimized preservation solution, mimicking the normal environment for the endothelium.

ELIGIBILITY:
Inclusion Criteria recipient:

* Age ≥18 years
* Signed informed consent form
* Listed for heart transplantation

Inclusion criteria donor:

* Age ≥18 and ≤70 years
* Accepted as heart donor by the transplant team
* (Research consent from the donor if required in country)

Exclusion Criteria recipient:

* Previous solid organ transplantation
* Grown-up congenital heart disease (GUCH)
* Kidney failure eGFR<40 at listing, calculated by CDK-EPI Creatinine, or ultrafiltration or dialysis or rapidly deteriorating kidney function due to a diagnosed renal disease
* Coagulopathy due to known hepatic disease or heparin induced thrombocytopenia
* Subject diagnosed with Systemic Lupus Erythematous, sarcoidosis or amyloidosis
* Known ongoing septicemia defined as positive blood culture immediately prior to the transplant (including with a durable VAD)
* Incompatible blood group
* Not able to understand the information provided during the informed consent procedure
* Combined organ transplantation candidates
* Subject already enrolled in another transplant related intervention study
* Subjects under pre-transplant desensitization protocol (including plasma exchange in conjunction with the transplant surgery)
* Mechanical circulatory support pre-transplantation (except durable Left ventricular assist device or Intra-aortic balloon pump)

Exclusion criteria donor:

* Previous sternotomy
* DCD hearts

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2020-11-25 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
30 days mortality and 30 days graft dysfunction | 30 days
  The Primary End-Point is defined as time-to-first-event of cardiac related death, moderate or severe primary graft dysfunction of the left ventricle or primary graft dysfunction of the right ventricle (according to Kobashigawa et al., 2014), acute cellular rejection ≥2R (according to Stewart et al., 2005) or graft failure (use of mechanical circulatory support or retransplantation) within 30 days.

SECONDARY OUTCOMES:
1 year mortality and 1 year graft dysfunction | 1 year
  The key secondary endpoint is defined as time-to-first-event of either any cause of death, moderate or severe PGD-LV or PGD-RV (according to Kobashigawa et al., 2014), acute cellular rejection ≥2R (according to Stewart et al., 2005) or graft failure (use of mechanical circulatory support or retransplantation) or CAV ≥ 1 (according to Mehra, 2010) within 12 months.
30 days and 1 year mortality and graft dysfunction | 30 days and 1 year
  The individual variables included in the composite primary endpoint at 30 days and 1 year analyzed as time-to-first-event.
CKMB | 3 days
  Creatine kinase MB (CKMB) at 6 ±2 h, 24 ±6 h, 48±6 h and 72±6 h after cross clamp removal
TnI | 3 days
  Tropinin I (TnI) at 6 ±2 h, 24 ±6 h, 48±6 h and 72±6 h after cross clamp removal
ProBNP | 3 days
  Pro Brain Natriuretic Protein (ProBNP) at 6 ±2 h, 24 ±6 h, 48±6 h and 72±6 h after cross clamp removal
Stay in ICU | 1 year
  Length of Stay at Intensive Care Unit, reported as number of days
Cardiac Transplant Events | 1 year
  Incidence of Major Adverse Cardiac Transplant Events
Postoperative use of mechanical circulatory support | 1 year
  Incidence of use of postoperative mechanical circulatory support, reported as number of days
Postoperative duration of mechanical circulatory support | 1 year
  Duration of use of postoperative mechanical circulatory support, reported as number of days
Overall success/failure 30 days | 30 days
  Success is defined as a recipient that are transplanted and alive at 30 days without any of the complication in the primary endpoint before 30 days.
Overall success/failure 1 year | 1 year
  Success is defined as a recipient that are transplanted and alive at 1 year without any of the complication given in key secondary endpoint before 1 year.
ECHO data (Left ventricular ejection fraction) | 24 hours
  ECHO data with Left ventricular ejection fraction in percentage within 24 hours after transplantation
ECHO data (Left ventricular ejection fraction) | 1 week
  ECHO data with Left ventricular ejection fraction in percentage 1 week after transplantation
ECHO data (Left ventricular ejection fraction) | 6 months
  ECHO data with Left ventricular ejection fraction in percentage 6 months after transplantation
ECHO data (Left ventricular ejection fraction) | 1 year
  ECHO data with Left ventricular ejection fraction in percentage 1 year after transplantation
ECHO data (Right ventricular ejection fraction) | 24 hours
  ECHO data with Right ventricular ejection fraction in percentage within 24 hours after transplantation
ECHO data (Right ventricular ejection fraction) | 1 week
  ECHO data with Right ventricular ejection fraction in percentage 1 week after transplantation
ECHO data (Right ventricular ejection fraction) | 6 months
  ECHO data with Right ventricular ejection fraction in percentage 6 months after transplantation
ECHO data (Right ventricular ejection fraction) | 1 year
  ECHO data with Right ventricular ejection fraction in percentage 1 year after transplantation
ECHO data (Tricuspid annular plane systolic excursion) | 24 hours
  ECHO data with Tricuspid annular plane systolic excursion (TAPSE) in mm within 24 hours after transplantation
ECHO data (Tricuspid annular plane systolic excursion) | 1 week
  ECHO data with Tricuspid annular plane systolic excursion (TAPSE) in mm 1 week after transplantation
ECHO data (Tricuspid annular plane systolic excursion) | 6 months
  ECHO data with Tricuspid annular plane systolic excursion (TAPSE) in mm 6 months after transplantation
ECHO data (Tricuspid annular plane systolic excursion) | 1 year
  ECHO data with Tricuspid annular plane systolic excursion (TAPSE) in mm 1 year after transplantation

OTHER OUTCOMES:
Serious adverse device effects | 1 year
  Incidence of any serious adverse device effects.
Adverse device effects | 1 year
  Incidence of any adverse device effects
Device dysfunction resulting in loss of transplantable heart | 12 hours
  Number of transplantable hearts lost due to device dysfunction
Intra operative details; duration of ECC | 12 hours
  Duration of ECC in minutes
Intra operative details; duration of cross clamp | 12 hours
  Duration of cross clamp in minutes
Intra operative details; duration of surgery | 12 hours
  Duration of surgery in minutes
Intra operative details; attempts to wean off ECC | 12 hours
  Number of attempts to wean off ECC
Intra operative details; need for inotropic support | 12 hours
  Need for inotropic support (inotropic score)
Intra operative details; need for pulmonary vasodilator | 12 hours
  Need for pulmonary vasodilator
Intra operative details; defibrillations | 12 hours
  Number of defibrillations
Intra operative details; arryhythmias | 12 hours
  Occurence of arryhythmias
Intra operative details; conduction abnormalities | 12 hours
  Number of conduction abnormalities
Intra operative details; Left ventricular ejection fraction (LVEF) | 12 hours
  LVEF in percentage
Intra operative details; Right ventricular ejection fraction (RVEF) | 12 hours
  RVEF in percentage
Intra operative details; Mitral valve regurgitations | 12 hours
  Grade of mitral valve regurgitations
Intra operative details; Tricuspid valve regurgitations | 12 hours
  Occurence of tricuspid vavle regurgitations
Arterial blood gas lactate | 6 hours
  Arterial blood gas lactate at 6 hours
Arterial blood gas lactate | 24 hours
  Arterial blood gas lactate at 24 hours
Pro-BNP during follow up | 1 year
  Pro-BNP at predefined time points during follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Filip Rega, MD, PhD, Principal Investigator — UZ Leuven
Locations (15):
- Allgemeines Krankenhaus der Stadt Wien, Vienna, Austria
- UZ Leuven, Leuven, Flemish Brabant, Belgium
- France (2):
  - Institut de cardiologie, Chirurgie thoracique et cardiovasculaire La Pitié Salpetrière, Paris, Paris Cedex
  - Hôpital Bichat Claude-Bernard, Paris
- Germany (5):
  - Klinikum der Universität München, München, Bavaria
  - Deutschen Herzzentrum Berlin, Berlin, Brandenburg
  - Universitätsklinik der Ruhr-Universität Bochum, Bad Oeynhausen
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Hannover Medical School, Hanover
- Azienda osedalaria di Padova, Padua, Padova PD, Italy
- Hospital Puerto de Hierro, Madrid, Majadahonda Madrid, Spain
- Sahlgrenska University Hospital, Gothenburg, Västra Götalands Regionen, Sweden
- United Kingdom (3):
  - Freeman Hospital, Newcastle, Newcastle upon Tyne
  - Queen Elisabeth Hospital, Birmingham
  - Royal Papworth Hospital, Cambridge

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rega F, Lebreton G, Para M, Michel S, Schramm R, Begot E, Vandendriessche K, Kamla C, Gerosa G, Berman M, Boeken U, Clark S, Ranasinghe A, Ius F, Forteza A, Pivodic A, Hennig F, Guenther S, Zuckermann A, Knosalla C, Dellgren G, Wallinder A; NIHP2019 investigators. Hypothermic oxygenated perfusion of the donor heart in heart transplantation: the short-term outcome from a randomised, controlled, open-label, multicentre clinical trial. Lancet. 2024 Aug 17;404(10453):670-682. doi: 10.1016/S0140-6736(24)01078-X. PMID 39153817
- [Derived] Brouckaert J, Dellgren G, Wallinder A, Rega F. Non-ischaemic preservation of the donor heart in heart transplantation: protocol design and rationale for a randomised, controlled, multicentre clinical trial across eight European countries. BMJ Open. 2023 Dec 28;13(12):e073729. doi: 10.1136/bmjopen-2023-073729. PMID 38154894